CLINICAL TRIAL: NCT06555978
Title: Ageing BIOmarker Study in Singaporeans (ABIOS)
Brief Title: Ageing BIOmarker Study in Singaporeans
Acronym: ABIOS
Status: Active, not recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Andrea Maier, Oon Chiew Seng Professor in Medicine, Healthy Ageing and Dementia Research, National University of Singapore
Other Study IDs: NHG-DSRB-2019-00388
Record Dates: First submitted 2024-08-08; First posted 2024-08-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy Aging; Biological Aging; Lifestyle Factors
Keywords: Aging; Biological Clocks; DNA methylation; Geroscience; Lifestyle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (serum, plasma, buffy, peripheral blood mononuclear cells), saliva (whole), and stool (whole) samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Singaporean adults: Adults greater than 21 years of age living in Singapore of Chinese, Malay, or Indian ethnicity.

SUMMARY:
The Ageing BIOmarker Study in Singaporeans (ABIOS) aims to understand the biological aging processes and how they affect health among people in Singapore. As people grow older, their risk of developing chronic diseases increases. This study aims to better understand the biological changes that come with age, particularly in three major ethnic groups: Chinese, Malay, and Indian adults over 21 years old. By examining a range of health indicators such as DNA methylation, inflammation, metabolism, cardiovascular health, physical function, and physical activity (i.e., molecular, physiological, and digital biomarkers of ageing), the study seeks to identify how ethnicity, lifestyle, and socioeconomic factors influence ageing. This unique study focuses on an all-Asian population, aiming to enhance our understanding of healthy aging across different ethnic groups.

DETAILED DESCRIPTION:
Biological ageing is the primary driver of age-associated chronic diseases in older adults. Asian populations have been underrepresented in studies developing biological age predictors and understanding age-related diseases. Thus, the Ageing BIOmarker Study in Singaporeans (ABIOS) aims to characterise the biomarkers of ageing in Singaporeans, exploring associations between molecular, physiological, and digital biomarkers of ageing.

This is a single-centre, cross-sectional study that recruits healthy community-dwelling adults (≥ 21 years) from three different ethnic groups (Chinese, Malay, and Indian). Molecular biomarkers of ageing include a multi-omics approach, such as DNA methylation and metabolic and inflammatory parameters in blood, saliva, and stool. Physiological biomarkers of ageing include bone density, body composition, skin autofluorescence, arterial stiffness, physical performance (e.g., muscle strength and flexibility), cognition, and nutritional status. Digital biomarkers of ageing include three-dimensional facial morphology and objective physical activity. Additional factors such as habitual physical activity, dietary patterns, and medical history are also examined. The associations between the molecular, physiological, and digital phenotypes will be explored.

By examining diverse age-related biomarkers, clinical indicators, and lifestyle factors, ABIOS will offer unique insights into the ageing process within these ethnic groups to develop health policies and interventions for promoting healthy ageing in an all-Asian population.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years of age
* Chinese, Malay, or Indian and has lived in Singapore for at least 5 consecutive years
* Apparently healthy and non-smokers
* Having only 1 condition (if ≥45 and <65 years) or any condition (if ≥65 years), and all conditions were medication-controlled (if any):

  * Hypertension
  * Hyperlipidemia
  * Hyperglycemia
  * Osteopenia/osteoporosis
  * Osteoarthritis
  * Type 2 diabetes

Exclusion Criteria:

* Body mass index (BMI) ≥30 kg/m^2
* Pre-existing or history of major cardiovascular disease (e.g., coronary artery disease, heart failure, stroke, peripheral vascular disease)
* Any metal implants (excluding dental implants) in the body
* Pre-existing or history of cancer or chronic obstructive pulmonary disease (COPD)
* Pregnant women or planning pregnancy in the next 6-12 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 21 years of age or greater who has lived in Singapore for at least 5 consecutive years and is of Chinese, Malay, or Indian ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
blood DNA methylation | Baseline
  DNA methylation ageing clock, years

SECONDARY OUTCOMES:
Carotid-femoral Pulse Wave Velocity | Baseline
  Arterial stiffness measured by pulse wave velocity, m/s
Handgrip strength | Baseline
  Handgrip strength measured by dynamometer, kg
8-repetition maximal strength | Baseline
  Lower body strength measured by maximum weight for 8 leg extension repetitions, kg
Skin autofluorescence | Baseline
  Skin autofluorescence measured by advanced glycation end products
Objective physical activity | Baseline
  Objective physical activity measured by an activity tracking monitor
Facial age | Baseline
  Facial ageing clock based on 3D face morphometry, years
Complete red blood cell (RBC) count | Baseline
  Clinical blood parameters, RBC x 10^12/L
Total white blood cell (WBC) count | Baseline
  Clinical blood parameters, WBC x 10^9/L
Total cholesterol | Baseline
  Lipid profile panel, mmol/L
HDL cholesterol | Baseline
  Lipid profile panel, mmol/L
LDL cholesterol | Baseline
  Lipid profile panel, mmol/L
Triglycerides | Baseline
  Lipid profile panel, mmol/L
Fasting blood glucose | Baseline
  Clinical blood parameters, mmol/L
Total protein | Baseline
  Liver profile panel, mmol/L
Total bilirubin | Baseline
  Liver profile panel, umol/L
Alkaline phosphatase (ALP) | Baseline
  Clinical blood parameters, U/L
Insulin | Baseline
  Clinical blood parameters, Roche immunoassay, mU/L
HbA1c | Baseline
  Clinical blood parameters, %

OTHER OUTCOMES:
Blood pressure | Baseline
  Central and brachial blood pressure measurements, mmHg
Waist-to-hip ratio | Baseline
  Waist-to-hip circumference ratio
Bone mineral density | Baseline
  Bone mineral density measured by DEXA scan, g/cm^2
Fat-free mass | Baseline
  Fat-free mass measured by DEXA scan, kg
Fat mass | Baseline
  Fat mass measured by DEXA scan, kg
Arm curl repetitions | Baseline
  Number of arm curl repetitions at a certain weight in 30 seconds
Backscratch test | Baseline
  Backscratch test to assess upper body flexibility, distance between fingers in cm
Sit-to-stand repeitions | Baseline
  Number of chair sit-to-stand repetitions in 30 seconds
4-metre walk | Baseline
  Time it takes for the participant to walk 4 metres, seconds
Habitual physical activity | Baseline
  Habitual physical activity patterns reflected by the Global Physical Activity Questionnaire
Cognitive function | Baseline
  Cognitive function test assessed by the Montreal Cognitive Assessment (MoCA)
Frailty | Baseline
  Frailty assessed by the FRAIL scale (fatigue, resistance, aerobic capacity, illnesses, and loss of weight), with three categories: robust (score=0), prefrail (score=1-2), and frail (score=3-5)
Risk of malnutrition | Baseline
  Risk of malnutrition assessed by the Mini Nutritional Assessment (MNA), with three categories: malnourished (0-7 points), at risk of malnutrition (8-11 points), normal nutritional status (12-14 points)
Saliva DNA methylation status | Baseline
  DNA methylation ageing clock, years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Maier, MD, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Centre for Healthy Longevity at Alexandra Hospital, Singapore, Singapore